CLINICAL TRIAL: NCT01206725
Title: The Effect of Aerobic Interval Training on Cardiac Function in Patients With Diabetes Mellitus Type 2 and Diastolic Dysfunction
Brief Title: Exercise Study on Cardiac Function in Patients With Diabetes Mellitus Type 2 and Diastolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2009.365
Record Dates: First submitted 2010-09-06; First posted 2010-09-22 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Type 2
Keywords: Diabetes type 2; exercise; tissue Doppler velocity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- . Moderate Intensity Exercise Group (Other): Exercise equivalent to the current exercise guidelines. In total 210 minutes per week of continuous moderate intensity (70% HRmax) exercise. Home based training.
  Interventions: Other: Exercise
- Aerobic interval training (Other): Exercise equivalent to the current guidelines achieved through high-intensity interval training.The exercise starts with warming-up for 10-min at 70% of HRmax before performing 4x4min intervals at 90-95% of HRmax, with 3-min active recovery at 70% of HRmax between each interval, and a 5-min cool-down period, giving a total of 40-min.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 1. Moderate Intensity Exercise Group (ME). Exercise equivalent to the current exercise guidelines. In total 210 minutes per week of continuous moderate intensity (70% HRmax) exercise. Home based training.
  2. Aerobic interval training (AIT). Exercise equivalent to the current guidelines achieved through high-intensity interval training.The exercise starts with warming-up for 10-min at 70% of HRmax before performing 4x4min intervals at 90-95% of HRmax, with 3-min active recovery at 70% of HRmax between each interval, and a 5-min cool-down period, giving a total of 40-min.

SUMMARY:
The aim of the study is to compare the effects of aerobic interval training and the IDF recommendations on physical activity on cardiac function and CV risk factors in patients with diabetes. The hypothesis is that AIT more than MCT, will improve myocardial dysfunction in patients with subclinical LV disease, improve both endothelial function and VO2max and thus reducing CV risk factors and CV disease. HbA1c will be more stable.

The aims of this study are to address the exercise prescription recommendations for patients with (T2DM) who have subclinical heart disease. The prescription recommendations will be assessed by randomising T2DM patients with subclinical heart disease to one of the following 2 groups for 3 months followed by a 9 month home-based program:

Moderate Intensity Exercise Group (ME). Home exercise equivalent to the present exercise recommendations of the International Diabetes Federation.

Aerobic interval training (AIT). Exercise equivalent to the current guidelines achieved through high-intensity interval training.

DETAILED DESCRIPTION:
The investigators primary hypotheses are that in patients with type 2 diabetes and subclinical heart disease:

Moderate Intensity Exercise will:

Not significantly improve myocardial function compared to controls,

Despite significant improvement (compared to controls) in:

Glycaemic control (HbA1c) Cardiorespiratory fitness (VO2max) Body composition (DXA)

Aerobic Interval Training Group will:

Significantly improve myocardial function compared to controls,

Significantly improve (compared to moderate intensity exercise group):

Glycaemic control (HbA1c) Cardiorespiratory fitness (VO2max) Body composition (DXA)

ELIGIBILITY:
Inclusion Criteria:

* Patients 20-60 years with diagnose diabetes mellitus type 2 (without insulin) for less than 10 years and with diastolic dysfunction (E'<8), will be included.

Exclusion Criteria:

* Overt CV disease
* History of CAD
* Moderate to severe valvular disease (AI MI 3-4, AS peak gradient > 15 mmHg=2m/s)
* Atrial fibrillation or other severe arrhythmia
* Congenital heart disease
* Untreated hypertension >140/90
* LVH
* Retinopathy
* Neuropathy
* Micro or macroalbuminuria
* EF < 40%
* BMI >35
* Ischemia at exercise echocardiography
* Disease or disability making training difficult.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Early diastolic tissue velocity (e') | 3 months

SECONDARY OUTCOMES:
Early diastolic tissue velocity (e') | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte B Ingul, PhD, Principal Investigator — NTNU, Det medisinske fakultet, Institutt for sirkulasjon og bildediagnostikk
Locations (1):
- Institutt for sirkulasjon og bildediagnostikk, Det medisinske fakultet,NTNU, Postboks 8905, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Hollekim-Strand SM, Bjorgaas MR, Albrektsen G, Tjonna AE, Wisloff U, Ingul CB. High-intensity interval exercise effectively improves cardiac function in patients with type 2 diabetes mellitus and diastolic dysfunction: a randomized controlled trial. J Am Coll Cardiol. 2014 Oct 21;64(16):1758-60. doi: 10.1016/j.jacc.2014.07.971. No abstract available. PMID 25323267
- [Result] Mallard AR, Hollekim-Strand SM, Coombes JS, Ingul CB. Exercise intensity, redox homeostasis and inflammation in type 2 diabetes mellitus. J Sci Med Sport. 2017 Oct;20(10):893-898. doi: 10.1016/j.jsams.2017.03.014. Epub 2017 Mar 21. PMID 28392340
- [Result] Hollekim-Strand SM, Hoydahl SF, Follestad T, Dalen H, Bjorgaas MR, Wisloff U, Ingul CB. Exercise Training Normalizes Timing of Left Ventricular Untwist Rate, but Not Peak Untwist Rate, in Individuals with Type 2 Diabetes and Diastolic Dysfunction: A Pilot Study. J Am Soc Echocardiogr. 2016 May;29(5):421-430.e2. doi: 10.1016/j.echo.2016.01.005. Epub 2016 Mar 3. PMID 26948543
- [Derived] Mallard AR, Hollekim-Strand SM, Ingul CB, Coombes JS. High day-to-day and diurnal variability of oxidative stress and inflammation biomarkers in people with type 2 diabetes mellitus and healthy individuals. Redox Rep. 2020 Dec;25(1):64-69. doi: 10.1080/13510002.2020.1795587. PMID 32693740